CLINICAL TRIAL: NCT05829434
Title: Magrolimab Plus Intensive Chemotherapy in Newly Diagnosed "ELN 2022 Intermediate or Adverse-risk" AML or High Risk MDS Patients Intended to Undergo Allogeneic Stem Cell Transplantation, a Phase 2, Single-arm, Open-Label Study
Brief Title: Magrolimab Plus Intensive Chemotherapy in Newly Diagnosed AML or HR-MDS
Acronym: MAGROLIC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was stopped prematurely due to safety reasons
Sponsor: Uwe Platzbecker (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Uwe Platzbecker, Clinical professor, University of Leipzig
Organization: University of Leipzig (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAGROLIC; EU Trial Number (Other: 2022-502040-13-00)
Record Dates: First submitted 2023-03-22; First posted 2023-04-25 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Neoplasm
Keywords: AML; Hihg-risk MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — magrolimab; Daunorubicin; Cytarabine; CPX-351

STUDY DESIGN:
Intervention Model Description: Patients are either treated with CPX-351 or 7+3
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magrolimab + intensive chemotherapy (7+3) (Experimental): Patients will receive magrolimab in combination with "7+3"
  Interventions: Drug: Magrolimab; Drug: 7+3
- Magrolimab + intensive chemotherapy (CPX-351) (Experimental): Patients will receive magrolimab in combination with CPX-351
  Interventions: Drug: Magrolimab; Drug: CPX-351

INTERVENTIONS:
Drug: Magrolimab — Patients will receive magrolimab on day 1; 4: IV 1 mg/kg; day 8: IV 15 mg/kg; day 11, 15 and 22: IV 30 mg/kg (plus 30 mg/kg for 5 weeks weekly and then q2w until the end of consolidation)
  Other Names: Hu5F9-G4; GS-4721
Drug: 7+3 — Patients will receive during Induction cycle 1: cytarabine at 100 mg/m² on study days 1-7 as a continuous infusion over 22-24 hours and daunorubicin at 60 mg/m² on study days 3, 4, 5
  * optional during Induction cycle 2: cytarabine at 100 mg/m² on days 1-7 of the second induction cycle (i.e. study days 29-35) as a continuous infusion over 22-24 hours and daunorubicin at 60 mg/m² on days 3, 4, 5 of the second induction cycle (i.e. study days 31, 32, 33)
  * optional during Consolidation cycle: cytarabine at 1 g/m² administered on days 1, 3, 5 of each consolidation cycle as an infusion for 2 hours every 12 hours (for patients < 60 years up to 3 CONS cycles and for patients ≥ 60 years up to 2 CONS cycles)
  Other Names: Daunorubicine and Cytarabine
  Arms: Magrolimab + intensive chemotherapy (7+3)
Drug: CPX-351 — Patients will receive during Induction cycle 1: CPX-351 with daunorubicin 44 mg/m² and cytarabine 100 mg/m² on days 1, 3, 5
  * optional during Induction cycle 2: CPX-351 with daunorubicin 44 mg/m² and cytarabine 100 mg/m² on days 29 + 30
  * optional during Consolidation cycle: CPX-351 with daunorubicin 29 mg/m² and cytarabine 65 mg/m² on days 1, 3
  Other Names: Vyxeos®
  Arms: Magrolimab + intensive chemotherapy (CPX-351)

SUMMARY:
Use of magrolimab in combination with standard intensive chemotherapy ("7+3" or CPX-351) in newly diagnosed "ELN 2022 intermediate or adverse-risk" AML or high risk MDS patients, who intend to undergo allogeneic stem cell transplantation

DETAILED DESCRIPTION:
Patients will receive magrolimab in combination with "7+3" or CPX-351 at:

* Day 1, 4: IV 1 mg/kg
* Day 8: IV 15 mg/kg
* Day 11, 15 and 22: IV 30 mg/kg
* Followed by weekly doses for 5 weeks and then q2w until the end of consolidation

If "7+3":

* Induction cycle 1 (IND 1):
* Cytarabine at 100 mg/m² on study days 1-7 as a continuous infusion over 22-24 hours
* Daunorubicin at 60 mg/m² on study days 3, 4, 5
* Induction cycle 2 (IND 2, optional):
* Cytarabine at 100 mg/m² on days 1-7 of the second induction cycle (i.e. study days 29-35) as a continuous infusion over 22-24 hours
* Daunorubicin at 60 mg/m² on days 3, 4, 5 of the second induction cycle (i.e. study days 31, 32, 33)
* Consolidation cycle (CONS, optional):
* Cytarabine at 1 g/m² administered on days 1, 3, 5 of each consolidation cycle as an infusion for 2 hours every 12 hours (for patients < 60 years up to 3 CONS cycles and for patients ≥ 60 years up to 2 CONS cycles)

If CPX-351:

* Induction cycle 1 (IND 1): CPX-351 (fixed combination daunorubicin 44 mg/m² and cytarabine 100 mg/m²) days 1, 3, 5
* Induction cycle 2 (IND 2, optional): CPX-351 (fixed combination daunorubicin 44 mg/m² and cytarabine 100 mg/m²) days 1, 3 (i.e. study days 29, 30)
* Consolidation cycle 1 (CONS, optional): CPX-351 (fixed combination daunorubicin 29 mg/m² and cytarabine 65 mg/m²) days 1, 3

ELIGIBILITY:
Inclusion Criteria:

* AML or MDS-IB2 according to WHO 2022 criteria
* For both MDS and AML: "Intermediate" or "adverse risk" genetic changes according to ELN 2022 category
* Eligible for and intention to undergo intensive chemotherapy (IC) (CPX-351 or "7+3") followed by allogeneic HSCT, as judged by the investigator

Exclusion Criteria:

* Patients harboring a FLT3mut, regardless of FLT3-ITD or FLT3-TKD mutation status and intended to receive midostaurin during induction and consolidation
* Patients intended to receive gemtuzumab-ozogamicin during intensive chemotherapy
* Patient does not accept bone marrow sampling during screening, during and after the treatment
* Patient does not accept several blood samplings during screening, treatment and after the treatment
* Patients who are not eligible for standard intensive chemotherapy as assessed by the treating physician
* Previous anthracycline-containing chemotherapy (Exception: cumulative dose for 1 cycle of planned induction therapy (CPX-351 or "7+3") not reached)
* Any prior treatment for AML or MDS (except for hydroxyurea or treatment for low-risk MDS e.g. growth factors) or prior treatment with CD47 or SIRPα-targeting agents, including magrolimab
* Inadequate organ function as defined as any criterion in the list below:

  1. Congestive heart failure or documented cardiomyopathy with an EF ≤50%
  2. Documented pulmonary disease with DLCO ≤65% or FEV1 ≤65%, or dyspnea at rest or requiring oxygen, or any pleural neoplasm or uncontrolled lung neoplasm
  3. On dialysis and age older than 60 years or uncontrolled renal carcinoma
  4. Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) > 5× upper limit of normal (ULN) or liver cirrhosis Child B or C or any biliary tree carcinoma or uncontrolled liver carcinoma or acute viral hepatitis
  5. Bilirubin > 1.5× ULN, or 3.0× ULN and primarily unconjugated if patient has a documented history of Gilbert's syndrome or genetic equivalent
  6. Serum creatinine > 1.5× ULN or calculated glomerular filtration rate (GFR) < 40 mL/min/1.73 m²
* ECOG performance status of ≥ 3
* Medical conditions other than MDS-IB-2 or AML with an estimated life expectancy below 3 months
* Relapsed or primary refractory AML
* Acute promyelocytic leukemia
* Known severe cardiopulmonary disease (e.g., unstable angina, congestive heart failure with an EF ≤50%, myocardial infarction within 6 months prior to screening, symptomatic cardiomyopathy, clinically significant arrhythmia17, clinically significant pulmonary hypertension requiring pharmacologic therapy)
* Uncontrolled high blood pressure (i.e., systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg)18
* Known prolonged rate-corrected QT interval ≥ 500 msec, calculated according to Fridericia's formula
* Active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Known active Human Immunodeficiency Virus infection (HIV 1/2 antibodies) with detectable viral load
* Known active Hepatitis B (i.e., HBsAg reactive) or Hepatitis C (i.e., HCV RNA [qualitative] is detected).
* Major surgery within 14 days of registration or a scheduled surgery during study period, depending on investigator decision
* Known uncontrolled central nervous system (CNS) involvement of MDS-IB-2 or AML (assessment by lumbar puncture is not mandatory for screening)
* Diagnosis or treatment for another malignancy within 1 year before registration and currently not in complete remission
* Any evidence of residual disease of another malignancy
* Patients with uncontrolled coagulopathy or bleeding disorder
* History or current evidence of any condition, therapy, or laboratory abnormality that might the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Current or planned pregnancy or nursing women (negative urine or serum pregnancy test within 3 days prior to receiving study treatment is needed. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test must be performed.)
* Female patients of childbearing potential, who are not using or not willing to use one highly effective method and one additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).
* Male patients, who do not agree to use an adequate method of contraception, starting with the first dose of study therapy during the entire study treatment period and through 3 months after the last dose of study drug. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s).
* Age under 18 years at registration
* Subject is unable to understand the nature, scope, significance and consequences of this clinical trial or has no legal capacity
* Simultaneous participation in another interventional clinical trial or participation in any clinical trial involving administration of an investigational medicinal product within 30 days prior to MAGROLIC trial registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Best CR/CRi/CRh | Up to 28 days
  Analysis of best CR/CRi/CRh (taken into count: number of neutrophils, platelets and bone marrow blasts) to describe efficacy of magrolimab in combination with intensive chemotherapy

SECONDARY OUTCOMES:
Overall Survival | up to 28 months
  Analysis of overall survival, OS (Time from study inclusion until death from any cause)
Event Free Survival | up to 57 days
  Analysis of event free survival, EFS (Time from study inclusion until end of induction (after up to two induction chemotherapies), hematological relapse or death from any cause (whichever comes first))
Relapse Free Survival | up to 28 months
  Analysis of relapse free survival, RFS (only for patients achieving CR); Time from achievement of complete remission until hematological relapse or death from any cause (whichever comes first)
Rate of allo HSCT | up to 28 days
  Rate of allogeneic hematopoietic stem cell transplantation, After induction cycle
Quality of life (EORTC QLQ-C30) | up to 4 months
  Evaluation according to EORTC QLQ-C30 Scoring Manual, Registration, during treatment and end of treatment
  To assess patient-reported quality of life during magrolimab treatment: 30 questions assessing the quality of life of oncology patients across 10 subscales will be analyzed. All subscales have a score range from 0 to 100 points.
  Function subscales: a higher score represents a higher quality of life. Symptoms subscales: higher score represents higher level of symptoms/problems, i.e., represents lower quality of life.
Quality of life (EQ-5D-5L) | up to 4 months
  Evaluation according to EQ-5D-5L User Guide, Registration, during treatment and end of treatment
  To assess patient-reported quality of life during magrolimab treatment within five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  Level 1 is coded as a '1', Level 2 is coded as a '2' and so on. Higher levels indicate lower quality of life..
Rate and severity of adverse events | up to 4 months
  Rate and severity of adverse events for patients treated with magrolimab and induction chemotherapy (Start of treatment up to end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof. Dr., Principal Investigator — University of Leipzig

IPD SHARING:
Plan to Share IPD: No